CLINICAL TRIAL: NCT03843333
Title: Feasibility of a CHW Intervention for Functional Decline in Rural Older Adults
Brief Title: A Community Health Worker Program to Support Rural Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Central Vermont Medical Center (Unknown); Dartmouth College (Other); Dartmouth-Hitchcock Medical Center (Other); MaineHealth (Other); MaineGeneral Health (Other); Maine-Dartmouth Family Medicine Residency (Unknown); Dartmouth SYNERGY Clinical and Translational Science Institute (Unknown); Northern New England Clinical and Translational Research Network (Unknown)
Responsible Party: Principal Investigator, Michael LaMantia, Section Head, Geriatric Medicine, Larner College of Medicine, University of Vermont
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-0685
Record Dates: First submitted 2019-02-07; First posted 2019-02-18 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Frail Elderly; Cognitive Impairment; Mobility Limitation; Depressive Symptoms
Keywords: Functional decline; Older adult; Community health workers; Cognitive impairment; Mobility limitation; Depressive symptoms; Rural; Primary care
MeSH Terms: conditions — Cognitive Dysfunction; Mobility Limitation; Depression

STUDY DESIGN:
Intervention Model Description: 24 participants at two intervention sites (n = 12 participants per site) will be compared with 24 participants at an enhanced usual care comparison site. We will also conduct qualitative interviews with 16 clinical staff and community health workers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHW Intervention (Experimental): CHWs will deliver three intervention components (Tai Ji Quan: Moving for Better Balance, Behavioral Activation, and Resource Navigation) to all participants at intervention sites over a 6-month period.
  Interventions: Behavioral: Tai Ji Quan: Moving for Better Balance; Behavioral: Behavioral Activation; Other: Resource Navigation
- Enhanced Usual Care (Active Comparator): Comparison participants will receive a guide on community resources for older adults, and assistance from the research team in making initial connections to resources if desired.
  Interventions: Other: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Tai Ji Quan: Moving for Better Balance — TJQMBB is an evidence-based, Centers for Disease Control and Prevention (CDC)-recommended, group falls prevention program based in Tai Chi that has been shown to reduce falls risk, improve physical function, and improve cognition. The program is delivered in 1-hour sessions twice weekly over 24 weeks, with the first 12 weeks spent learning the basic Tai Ji Quan forms and the second 12 weeks focused on variations in practice that progressively increase physical and cognitive demands. A physical therapist at Dartmouth is an authorized TJQMBB trainer and will train the CHWs to deliver the intervention and provide remote supervision monthly.
  Arms: CHW Intervention
Behavioral: Behavioral Activation — BA is a brief intervention for depressive symptoms that focuses on engagement in positively-reinforcing activities and decreasing activity avoidance. CHWs will be trained by Dartmouth psychologists to deliver a brief behavioral activation program to encourage participants to increase their involvement in meaningful activities. BA will be delivered in one-hour sessions in the home every other week for 12 weeks. Supervision will be provided remotely on a weekly basis.
  Arms: CHW Intervention
Other: Resource Navigation — CHWs will assess participants' unmet psychosocial needs and assist them in identifying and connecting them with resources to address these needs.Types of assistance may include identifying transportation services, assisting with applications for benefits, linking participants to Meals on Wheels and other local food resources, and connecting participants to community programs for older adults. We expect that participant needs and services delivered will vary and acknowledge that this intervention component will not be standardized due to the nature of this work.
  Arms: CHW Intervention
Other: Enhanced Usual Care — Comparison participants will receive a detailed resource guide on community supports for older adults. The research team will facilitate referrals to local resources (e.g. the Dartmouth Aging Resource Center) if desired by participants. Data from research assessments of cognition, depressive symptoms, mobility, and functional status will be provided to the primary care team for follow-up and intervention as needed.
  Arms: Enhanced Usual Care

SUMMARY:
This study will investigate an intervention delivered by community health workers for older adults with signs of cognitive impairment, mobility loss, and depression in the rural primary care setting.

DETAILED DESCRIPTION:
The population of the United States is aging rapidly, and the populations of Vermont (VT), New Hampshire (NH), and Maine (ME) are among the oldest in the nation. There is a need to develop and disseminate interventions to prevent functional decline in older adults, defined as difficulty completing daily activities independently. Cognitive impairment, depressive symptoms, and mobility loss are three common syndromes identified in primary care that contribute to functional decline in older adults. Evidence-based interventions can address early stages of these three conditions; however older adults in rural communities may have particular difficulty accessing interventions due to limited health and social services. Community health workers (CHWs) offer a potential strategy to address gaps in care and deliver interventions to vulnerable older adults in rural communities.

The overarching goal of this study is to conduct a pilot investigation of a CHW-delivered intervention to slow progression of functional decline among at-risk older adults. Using qualitative and quantitative methods, this pilot study will: 1) Evaluate whether a multicomponent intervention delivered by CHWs for rural older adults at risk for functional decline is feasible to deliver and acceptable to older adults and their primary care teams; and 2) Explore the effectiveness of combined Tai Ji Quan: Moving for Better Balance (TJQMBB), behavioral activation (BA), and resource navigation in slowing functional decline among older adults with co-occurring early impairments in cognition, mood, and mobility.

Older adults who are at high risk for functional decline will be recruited from partnering primary care sites (two intervention sites in VT and ME, and one comparison site in NH) based on results from the Medicare Annual Wellness Visit (AWV), which incorporates screening for cognitive impairment, depression, and falls risk, as well as provider referral and chart review. CHWs will be trained to deliver a 6-month intervention incorporating two evidence-based interventions that target cognition, depressive symptoms, and mobility (TJQMBB and behavioral activation), and resource navigation to address unmet social needs that may create barriers. Feasibility, acceptability, and potential effectiveness will be assessed through a combination of qualitative interviews, standardized questionnaires, physical measurements, and surveys.

ELIGIBILITY:
Inclusion Criteria:

* Age 65 or greater
* Positive for at least 2 of the following: 1) PHQ-2 score ≥2 or PHQ-9 score ≥5; 2) Mini-Cog score <4 or MoCA score <26 or Six-item screener with ≥2 errors; 3) "Yes" response to any of 3 falls risk screening questions or Timed Up and Go time 12 seconds or higher

Exclusion Criteria:

* Active suicidal ideation
* PHQ-9 score >14
* MoCA score <19
* Inability to ambulate (use of an assistive device is acceptable)
* Inability to stand steadily in a stationary position without support
* Physician objection to participation due to medical, psychological, or other concerns
* Inability to speak and understand English
* Lack of capacity to provide informed consent as determined by the University of California, San Diego Brief Assessment of Capacity to Consent (UBACC)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Change in functional status from as measured by the Complete Activities of Daily Living Section of the Older Americans' Resources and Services (OARS) Multidimensional Functional Assessment Questionnaire | Baseline, 3, 6, and 9 months.
  A 14-item self-report measure of independence in performing Activities of Daily Living (ADLs) and Instrumental Activities of Daily Living (IADLs). Scores range from 0-28 with a score of 0 indicating complete dependence in activities and 28 indicating complete independence. ADL and IADL subscales each have 7 items scored from 0-14 which are summed to calculate the total score.

SECONDARY OUTCOMES:
Change in cognitive function as measured by the Montreal Cognitive Assessment (MoCA) | Baseline, 3, 6, and 9 months.
  A brief interviewer-delivered cognitive assessment that assesses visuospatial/executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation. Scores range from 0-30 with a high score of 26-30 indicating normal cognitive function.
Change in depressive symptom severity as measured by the Patient Health Questionnaire (PHQ-9) | Baseline, 3, 6, and 9 months.
  A 9-item self-report measure of severity of depressive symptoms. Scores range from 0-27 with 0-4 indicating no or minimal depression, 5-9 indicating mild depression, 10-14 indicating moderate depression, 15-19 indicating moderately severe depression, and 20-27 indicating severe depression.
Change in mobility as measured by the Timed Up and Go (TUG) | Baseline, 3, 6, and 9 months.
  Time (in seconds) to rise from a chair, walk 10 feet, and return to seated position in chair. A time of 12 seconds of higher indicates falls risk.
Change in mobility as measured by the 30-Second Chair Stand | Baseline, 3, 6, and 9 months.
  Number of times participant is able to rise to a standing position from a chair in 30 seconds. Age and gender-specific cutoffs are used to determine falls risk (e.g. scores less than 12 for men and less than 11 for women are considered abnormal for age 65-69).

OTHER OUTCOMES:
Change in handgrip strength | Baseline, 3, 6, and 9 months.
  Measured grip strength using a handheld Jamar dynamometer.
Change in falls frequency. | Baseline, 3, 6, and 9 months.
  Self-reported number of falls in the past 3 months.
Change in social support as measured by the Duke Social Support Index | Baseline, 3, 6, and 9 months.
  11-item self-report measure of social support for the elderly, with scores ranging from 11-33 (low social support to high social support). Social Interaction (range 4-12) and Subjective Social Support (range 7-21) subscales are totaled for the overall score.
Change in self-reported general health status as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Global Health Scale v1.2. | Baseline, 3, 6, and 9 months.
  10-item self-report measure of global physical and mental health status. Raw summed scores of 4-20 (higher scores indicates better functioning) for physical and mental health subscales are converted to standardized T-scores each with a mean of 50.
Number and type of social needs and community resources used as measured by a checklist | Baseline, 3, 6, and 9 months.
  Brief checklist to assess psychosocial needs (e.g. financial concerns, transportation problems, food insecurity) and types of community resources used in the past 3 months.
Health care utilization as measured by past 3 month Emergency Department (ED) visits | Baseline, 3, 6, and 9 months.
  Number of ED visits in the past 3 months.
Health care utilization as measured by past 3 month hospitalizations | Baseline, 3, 6, and 9 months.
  Number of hospitalizations in the past 3 months.
Health care utilization as measured by past 3 month long-term care placements | Baseline, 3, 6, and 9 months.
  Number of long-term care placements in the past 3 months.
Feasibility and acceptability as determined by qualitative interviews | At completion of study, approximately 9 months.
  Semi-structured interviews will be conducted with participants, clinical staff, and CHWs and will undergo thematic analysis.
Fidelity of TJQMBB as measured by fidelity checklist | At completion of TJQMBB phase of intervention, approximately 6 months.
  Percent of intervention sessions with fidelity based on checklist of required components.
Fidelity of BA as measured by fidelity checklist | At completion of BA phase of intervention, approximately 3 months
  Percent of intervention sessions with fidelity based on checklist of required components.
Acceptability of the intervention as measured by satisfaction survey | At completion of intervention phase, approximately 6 months.
  Percent of participant satisfaction surveys with positive ratings.
Acceptability of intervention as measured by completion of TJQMBB sessions | At completion of TJQMBB phase of intervention, approximately 6 months.
  Percent of scheduled TJQMBB sessions attended by participants.
Acceptability of intervention as measured by completion of BA sessions | At completion of BA phase of intervention, approximately 3 months.
  Percent of scheduled BA sessions completed by participants.
Feasibility of recruitment | At recruitment completion, approximately 3 months.
  Ability to recruit n = 24 intervention and n = 24 comparison participants.
Retention | At study completion, approximately 9 months.
  Percent of scheduled study assessment visits completed by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A LaMantia, MD, MPH, Principal Investigator — University of Vermont
Locations (3):
- United States (3):
  - Maine Dartmouth Geriatric Medicine, Augusta, Maine
  - Dartmouth-Hitchcock Lyme, Lyme, New Hampshire
  - Integrative Family Medicine - Montpelier, Montpelier, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li F, Harmer P, Fisher KJ, McAuley E, Chaumeton N, Eckstrom E, Wilson NL. Tai Chi and fall reductions in older adults: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2005 Feb;60(2):187-94. doi: 10.1093/gerona/60.2.187. PMID 15814861
- [Background] Li F, Harmer P, Liu Y, Chou LS. Tai Ji Quan and global cognitive function in older adults with cognitive impairment: a pilot study. Arch Gerontol Geriatr. 2014 May-Jun;58(3):434-9. doi: 10.1016/j.archger.2013.12.003. Epub 2013 Dec 22. PMID 24398166
- [Background] Li F. Transforming traditional Tai Ji Quan techniques into integrative movement therapy-Tai Ji Quan: Moving for Better Balance. J Sport Health Sci. 2014 Mar 1;3(1):9-15. doi: 10.1016/j.jshs.2013.11.002. PMID 25126445
- [Background] Orgeta V, Brede J, Livingston G. Behavioural activation for depression in older people: systematic review and meta-analysis. Br J Psychiatry. 2017 Nov;211(5):274-279. doi: 10.1192/bjp.bp.117.205021. Epub 2017 Oct 5. PMID 28982660
- [Background] Lejuez CW, Hopko DR, Acierno R, Daughters SB, Pagoto SL. Ten year revision of the brief behavioral activation treatment for depression: revised treatment manual. Behav Modif. 2011 Mar;35(2):111-61. doi: 10.1177/0145445510390929. PMID 21324944
- [Background] Rosenthal EL, Brownstein JN, Rush CH, Hirsch GR, Willaert AM, Scott JR, Holderby LR, Fox DJ. Community health workers: part of the solution. Health Aff (Millwood). 2010 Jul;29(7):1338-42. doi: 10.1377/hlthaff.2010.0081. PMID 20606185
- [Background] Kim K, Choi JS, Choi E, Nieman CL, Joo JH, Lin FR, Gitlin LN, Han HR. Effects of Community-Based Health Worker Interventions to Improve Chronic Disease Management and Care Among Vulnerable Populations: A Systematic Review. Am J Public Health. 2016 Apr;106(4):e3-e28. doi: 10.2105/AJPH.2015.302987. Epub 2016 Feb 18. PMID 26890177
- [Background] Barnett ML, Gonzalez A, Miranda J, Chavira DA, Lau AS. Mobilizing Community Health Workers to Address Mental Health Disparities for Underserved Populations: A Systematic Review. Adm Policy Ment Health. 2018 Mar;45(2):195-211. doi: 10.1007/s10488-017-0815-0. PMID 28730278
- See also: American Public Health Association Policy Statement on Community Health Workers — https://www.apha.org/policies-and-advocacy/public-health-policy-statements/policy-database/2014/07/09/14/19/support-for-community-health-workers-to-increase-health-access-and-to-reduce-health-inequities
- See also: Web site for Tai Ji Quan: Moving for Better Balance program — https://tjqmbb.org/